CLINICAL TRIAL: NCT01344824
Title: A Multicenter Phase II Trial of Carboplatin, Pemetrexed, and Bevacizumab Followed By Pemetrexed and Bevacizumab Maintenance Therapy in Patients With a Light or Never Smoking History
Brief Title: Carboplatin, Pemetrexed Disodium, and Bevacizumab for Patients With Stage III or IV Non-Small Cell Lung Cancer Who Are Light/Never Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0825; P30CA016086 (NIH)
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Carboplatin; Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Trial (Other): Bevacizumab, Carboplatin, and Pemetrexed disodium, with option for second line erlotinib hydrochloride
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: erlotinib hydrochloride; Drug: pemetrexed disodium

INTERVENTIONS:
Biological: bevacizumab — 15 mg/kg once per 21 day cycle (up to 4 cycles).
  Other Names: Avastin
Drug: carboplatin — Area Under the Curve (AUC)=6, once every 21 day cycle (up to 4 cycles)
  Other Names: Paraplatin
Drug: erlotinib hydrochloride — 150mg, daily for 21 day cycle (up to 4 cycles)
  Other Names: Tarceva
Drug: pemetrexed disodium — 500 mg/m2 on day 1 of a 21 day cycle (up to 4 cycles)
  Other Names: ALIMTA

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Giving carboplatin and pemetrexed disodium together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving carboplatin and pemetrexed disodium together with bevacizumab works in treating patients with stage III or stage IV non-small cell lung cancer who are light or never smokers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the progression-free survival (PFS) of patients with advanced non-small cell lung cancer who are never or light smokers treated with carboplatin, pemetrexed disodium, and bevacizumab followed by pemetrexed disodium and bevacizumab maintenance therapy.

Secondary

* To estimate the overall survival (OS) of patients treated with this regimen.
* To estimate the toxicity of treatment using the NCI CTCAE version 3.0.
* To conduct an exploratory analysis of molecular markers, e.g., Kirsten rat sarcoma (KRAS) and epidermal growth factor receptor (EGFR) mutations, in patients with a never or light smoking history and to analyze any potential association with response, PFS, and OS.
* To assess response to second-line erlotinib hydrochloride therapy according to RECIST criteria.

OUTLINE: This is a multicenter study.

* First-line therapy: Patients receive pemetrexed disodium IV over 10 minutes, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients who achieve partial or complete response or have stable disease progress to maintenance therapy.
* Maintenance therapy: Patients receive pemetrexed disodium IV over 10 minutes and bevacizumab IV over 30 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients who experience disease progression or unacceptable toxicity may receive second-line therapy with erlotinib hydrochloride as part of standard-of-care treatment.

Tissue samples are collected at baseline for laboratory biomarker analysis.

After completion of maintenance therapy, patients are followed every 4 weeks for 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary lung carcinoma

  * Non-squamous histology
  * Advanced disease defined as stage IIIB disease with cytologically documented malignant pleural or pericardial effusion or stage IV disease
* Available pathology block or unstained slides from initial or subsequent diagnosis

  * Must have undergone ≥ 1 core biopsy
  * No patients whose diagnosis was made through a fine-needle aspirate
* No uncontrolled pleural effusions, ascites, or third-space fluid collections
* Meets 1 of the following criteria:

  * Non-smoker, defined as patients who smoked ≤ 100 cigarettes in their lifetime
  * Former light smoker, defined as patients who smoked between > 100 cigarettes AND ≤ 10 pack-years AND quit ≥ 1 year ago
* No known central nervous system disease, except for treated brain metastases meeting the following criteria:

  * No evidence of progression or hemorrhage after treatment
  * No ongoing requirement for dexamethasone as ascertained by clinical examination and brain imaging (MRI or CT scan) during the screening period
  * Stable doses of anticonvulsants are allowed
  * Treatment for brain metastases may include whole-brain radiotherapy, radiosurgery (gamma knife, LINAC, or equivalent), or a combination as deemed appropriate by the treating physician
  * No patients with central nervous system (CNS) metastases treated by neurosurgical resection
  * No brain biopsy within the past 3 months

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST/ALT) ≤ 2.5 times ULN
* Calculated creatinine clearance > 45 mL/min OR creatinine ≤ 1.5 times ULN
* Prothrombin time ≤ 1.5 times ULN
* Partial thromboplastin time ≤ ULN
* Urine protein:creatinine ratio ≤ 1.0
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Patients with a history of hypertension are eligible provided it is well controlled (BP < 150/100 mm Hg) on a stable regimen of antihypertensive therapy

  * No history of hypertensive crisis or hypertensive encephalopathy
* Able and compliant with folic acid and B12 supplementation
* Able to swallow tablets intact or dissolved in water
* No dysphagia or active gastrointestinal (GI) disease or disorder that alters GI motility or absorption
* No lack of integrity of the GI tract (e.g., a significant surgical resection of the stomach or small bowel)
* No abdominal fistula, GI perforation, or intraabdominal abscess within the past 6 months
* None of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure (NYHA class II-IV)
  * Cardiac arrhythmia
  * Psychiatric illness, social situations, or any other medical condition that would limit compliance with study requirements
* No myocardial infarction or other evidence of arterial thrombotic disease (angina) within the past 6 months
* No history of cerebral vascular accident or transient ischemic attack within the past 6 months
* No significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within the past 6 months
* No history of bleeding diathesis or coagulopathy
* No ongoing hemoptysis, defined as ≥ ½ teaspoon of bright red blood

  * Patients with procedure-related hemoptysis that has resolved post-procedure are eligible
* No serious nonhealing wound, ulcer, bone fracture, or significant traumatic injury within the past 28 days
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy

  * Patient must be chemotherapy naive
  * Prior neoadjuvant or adjuvant chemotherapy allowed provided it was completed ≥ 6 months ago
* No prior anti-vascular endothelial growth factor therapy
* At least 3 weeks since prior major surgery
* At least 1 week since prior radiotherapy
* More than 28 days since prior and no concurrent treatment with an investigational agent
* More than 7 days since prior core biopsy
* Concurrent daily treatment with aspirin or NSAIDs are eligible provided patients are able to interrupt NSAIDs 2 days before (5 days for long-acting NSAIDs), the day of, and for 2 days following the administration of pemetrexed disodium
* No concurrent treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix), and/or cilostazol (Pletal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-03; Primary Completion 2016-05-24 (Actual); Study Completion 2016-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Stinchcombe, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Mission Hospital, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - CCHC New Bern Cancer Care, New Bern, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiss JM, Villaruz LC, O'Brien J, Ivanova A, Lee C, Olson JG, Pollack G, Gorman R, Socinski MA, Stinchombe TE. Results of a Phase II Trial of Carboplatin, Pemetrexed, and Bevacizumab for the Treatment of Never or Former/Light Smoking Patients With Stage IV Non-Small Cell Lung Cancer. Clin Lung Cancer. 2016 Mar;17(2):128-32. doi: 10.1016/j.cllc.2015.12.006. Epub 2015 Dec 17. PMID 26774201
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from institutions including University of North Carolina Hospitals, University of Pittsburgh Medical Center, Mission Cancer Center, and New Bern Cancer Center.
Pre-assignment Details: From March 2010 to November 2013, 52 patients consented to treatment. 14 patients were consented and screened for eligibility but found ineligible.
Groups:
- Bevacizumab, Carboplatin, and Pemetrexed Disodium, With Option: Bevacizumab, Carboplatin, and Pemetrexed disodium, with option for second line erlotinib hydrochloride
  bevacizumab: 15 mg/kg once per 21 day cycle (up to 4 cycles).
  carboplatin: Area Under the Curve (AUC)=6, once every 21 day cycle (up to 4 cycles)
  erlotinib hydrochloride: 150mg, daily for 21 day cycle (up to 4 cycles)
  pemetrexed disodium: 500 mg/m2 on day 1 of a 21 day cycle (up to 4 cycles)
Period: Overall Study
Arm/Group | Bevacizumab, Carboplatin, and Pemetrexed Disodium, With Option
Started | 38
Completed | 1
Not Completed | 37
Not completed — Adverse Event | 15
Not completed — Withdrawal by Subject | 6
Not completed — Other complicating disease | 1
Not completed — Progression | 15

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 63.5 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 30
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 38
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale from 0-5 to describe a patient's level of functioning in terms of selfcare ability and activity level.
  0, Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    grade 0 | 18
    grade 1 | 14
    not performed | 6
Smoking Status [Count of Participants; unit: Participants]
  Never smoker | 24
  Former light smoker | 14
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 37
  Neuroendocrine carcinoma | 1
Previous erlotinib treatment [Count of Participants; unit: Participants] | 10
Mutation status [Count of Participants; unit: Participants]
  EGFR | 6
  KRAS | 5
  EML4/ALK | 0
  MET del14 | 1
  None (tested and no driver found) | 22
  Unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Documented radiographic response per Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by imaging: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. criteria each year, until subject death
Time Frame: 1400 days
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 38
months | 12.6 [8.0 to 30.5]

2. Secondary Outcome: Overall Survival
Description: Time of enrollment to date of death.
Time Frame: 1400 days
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Trial
Number analyzed (Participants) | 38
months | 20.3 [15.8 to 30.5]

3. Secondary Outcome: Subjects Experiencing Toxicity
Description: Toxicity will be evaluated using CTCAE criteria, version 3, all grade 3 and 4 events.
Time Frame: 90 days
Population: All patients who received treatment were evaluated
Measure: Number; unit: participants
Arm/Group | Bevacizumab, Carboplatin, and Pemetrexed Disodium, With Option
Number analyzed (Participants) | 38
participants
  Diarrhea | 3
  Dyspnea (shortness of breath) | 2
  Fatigue (asthenia, lethargy, malaise) | 6
  Hemoglobin | 6
  Hypertension | 6
  Leukocytes (total white blood cell count) | 2
  Lymphopenia | 4
  Nausea | 2
  Neutrophils/granulocytes (ANC/AGC) | 7
  Joint pain | 2
  Platelets | 2
  Vomiting | 2

ADVERSE EVENTS:
Time Frame: Five years from registration
Arm/Group | Single Arm Trial
All-Cause Mortality (participants affected / at risk) | 28/38
Serious Adverse Events (participants affected / at risk) | 14/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=38)
Ataxia (incoordination) (Nervous system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Extremity-lower (gait/walking) (General disorders) | 1
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Lung (pneumonia) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Kidney (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Rectum (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1
Infection with unknown ANC - Kidney (Infections and infestations) | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Pain - Pain NOS (General disorders) | 1
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 2
Syncope (fainting) (Nervous system disorders) | 1
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Trial (N=38)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
Alkaline phosphatase (Metabolism and nutrition disorders) | 3
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 7
Anorexia (Metabolism and nutrition disorders) | 6
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 9
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 1
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 2
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Creatinine (Metabolism and nutrition disorders) | 5
Dehydration (Gastrointestinal disorders) | 1
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 3
Diarrhea (Gastrointestinal disorders) | 8
Distension/bloating, abdominal (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 8
Dry eye syndrome (Eye disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7
Edema: head and neck (General disorders) | 1
Edema: limb (General disorders) | 7
Extremity-lower (gait/walking) (General disorders) | 2
Eyelid dysfunction (Eye disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 29
Febrile neutropenia(ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Blood and lymphatic system disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 5
Flu-like syndrome (General disorders) | 1
Flushing (Vascular disorders) | 1
Glomerular filtration rate (Renal and urinary disorders) | 2
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 11
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Hematoma (Vascular disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 19
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 2
Hemorrhage, pulmonary/upper respiratory - Bronchopulmonary NOS (Respiratory, thoracic and mediastinal disorders) | 4
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 8
Hemorrhage/Bleeding - Other (Specify, __) (Vascular disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 2
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 12
Hypotension (Vascular disorders) | 2
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Abdomen NOS (Infections and infestations) | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Lip/perioral (Infections and infestations) | 1
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Upper airway NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Bronchus (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Kidney (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Nose (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Pharynx (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Rectum (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Vagina (Infections and infestations) | 1
Infection with unknown ANC - Kidney (Infections and infestations) | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1
Infection with unknown ANC - Middle ear (otitis media) (Infections and infestations) | 1
Infection with unknown ANC - Oral cavity-gums (gingivitis) (Infections and infestations) | 1
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 1
Infection with unknown ANC - Upper airway NOS (Infections and infestations) | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1
INR (International Normalized Ratio of prothrombin time) (Investigations) | 1
Insomnia (Psychiatric disorders) | 3
Intra-operative injury - Extremity-upper (Injury, poisoning and procedural complications) | 1
Intra-operative Injury - Other (Specify, __) (Injury, poisoning and procedural complications) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 6
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3
Mood alteration - Depression (Psychiatric disorders) | 5
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 3
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Extraocular (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-lower (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 21
Neurology - Other (Specify, __) (Nervous system disorders) | 1
Neuropathy: cranial - CN II Vision (Nervous system disorders) | 1
Neuropathy: cranial - CN VIII Hearing and balance (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 10
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2
Otitis, external ear (non-infectious) (Ear and labyrinth disorders) | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 2
Pain - Bladder (Renal and urinary disorders) | 2
Pain - Bone (Musculoskeletal and connective tissue disorders) | 3
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 3
Pain - Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 3
Pain - Dental/teeth/peridontal (Gastrointestinal disorders) | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 6
Pain - Head/headache (Nervous system disorders) | 9
Pain - Intestine (Gastrointestinal disorders) | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 9
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1
Pain - Oral cavity (Gastrointestinal disorders) | 1
Pain - Other (Specify, __) (General disorders) | 3
Pain - Pain NOS (General disorders) | 3
Pain - Pelvis (Musculoskeletal and connective tissue disorders) | 1
Pain - Rectum (Gastrointestinal disorders) | 2
Pain - Sinus (Respiratory, thoracic and mediastinal disorders) | 2
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 3
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
Phlebitis (including superficial thrombosis) (Vascular disorders) | 2
Platelets (Blood and lymphatic system disorders) | 7
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4
PTT (Partial Thromboplastin Time) (Investigations) | 1
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5
Soft tissue necrosis - Extremity-upper (Musculoskeletal and connective tissue disorders) | 1
Supraventricular and nodal arrhythmia - Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 2
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1
Vision-blurred vision (Eye disorders) | 2
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 9
Watery eye (epiphora, tearing) (Eye disorders) | 3
Weight gain (Investigations) | 1
Weight loss (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No